CLINICAL TRIAL: NCT06840379
Title: Effects of Sertraline on C-Reactive Protein Serum Levels in Hemodialysis Patients Diagnosed with Depression
Brief Title: Effect of Sertraline on Inflammation in Hemodialysis Patients with Depression: a Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Amra Batool, Principal Investigator, Nishtar Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NishtarMU3
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Inflamation; Hemodialysis; End Stage Renal Disease on Hemodialysis (Diagnosis)
Keywords: Depression in Chronic Kidney Disease; Hemodialysis and Mental Health; Sertraline and Inflammation; C-Reactive Protein and Depression; Psychiatric Comorbidities in ESRD
MeSH Terms: conditions — Disease; Psychological Well-Being; Inflammation; Depression | interventions — Sertraline; Antidepressive Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sertraline Group (Experimental): Participants in this group will receive oral sertraline, starting at 25 mg/day, with titration up to 100 mg/day based on clinical response and tolerability over the 12-week study period.
  Interventions: Drug: Sertraline (Oral Antidepressant)
- Placebo Group (Placebo Comparator): Participants in this group will receive an identical placebo tablet orally, following the same dosing schedule as the sertraline group for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline (Oral Antidepressant) — * 25 mg/day sertraline, titrated up to 100 mg/day based on clinical response and tolerability.
  * Administered orally once daily for 12 weeks.
  * Used to assess its effects on C-reactive protein (CRP) levels and depressive symptoms in hemodialysis patients.
  Arms: Sertraline Group
Drug: Placebo — * Identical placebo tablet administered orally once daily for 12 weeks, following the same dosing schedule as the sertraline group.
  * Used to compare the effects of sertraline vs. placebo on CRP levels and depression severity in hemodialysis patients.
  Arms: Placebo Group

SUMMARY:
Depression is a common mental health condition among patients undergoing hemodialysis and is associated with a lower quality of life, poor treatment adherence, and worse overall health outcomes. Chronic inflammation, as measured by elevated C-reactive protein (CRP) levels, is frequently seen in these patients and contributes to an increased risk of cardiovascular disease, the leading cause of death in this population.

Sertraline, a widely used antidepressant, is effective in treating depression in hemodialysis patients and has been suggested to have anti-inflammatory properties. This study aims to evaluate whether sertraline can reduce inflammation, as measured by CRP levels, in hemodialysis patients diagnosed with depression.

This research is a randomized, double-blind, placebo-controlled trial conducted at Nishtar Hospital, Multan. A total of 62 adult hemodialysis patients with depression will be enrolled and randomly assigned to receive either sertraline or a placebo for 12 weeks.

Depression severity will be assessed using the Hamilton Depression Rating Scale (HAM-D), a widely used tool for measuring the severity of depressive symptoms. HAM-D scores will be recorded at baseline, at weeks 4, 8, and 12 to evaluate changes in depressive symptoms over time.

CRP levels will also be measured at baseline and after 12 weeks to determine whether sertraline reduces systemic inflammation in these patients.

The hypothesis of this study is that sertraline treatment will significantly lower CRP levels compared to a placebo, potentially providing dual benefits-improving mood and reducing inflammation-related health risks in hemodialysis patients. The findings of this study could help improve treatment strategies for depression and inflammation in individuals undergoing long-term dialysis.

DETAILED DESCRIPTION:
After obtaining ethical approval, eligible participants were recruited from the hemodialysis unit. The study purpose, procedures, risks, and benefits were explained, and written informed consent was obtained. Participants meeting inclusion criteria underwent baseline assessments, including demographic data, medical history, HAM-D scores, and blood sampling for CRP measurement. Participants were randomly assigned to receive either sertraline or placebo using a computer-generated randomization sequence. The sertraline group initially received 25 mg/day, titrated up to a maximum of 100 mg/day over 4 weeks based on clinical response and tolerability. The placebo group received identical-looking tablets. Participants were monitored for 12 weeks, with follow-up visits every 2 weeks. Adherence, side effects, and any changes in medical status were assessed at each visit. At the end of 12 weeks, final HAM-D scores were obtained, and blood samples were collected for CRP measurement. All data were recorded on a standardized form.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* On maintenance hemodialysis for at least 3 months
* Diagnosed with depression as per operational definition
* Stable on current medications for at least 4 weeks

Exclusion Criteria:

* Current use of antidepressants or anti-inflammatory drugs
* Active infection or inflammatory condition
* History of bipolar disorder or psychosis
* Pregnancy or breastfeeding
* Severe liver disease (Child-Pugh class C)
* Known hypersensitivity to sertraline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Serum C-Reactive Protein (CRP) Levels from Baseline to 12 Weeks | Baseline and Week 12
  The mean change in CRP levels (mg/L) from baseline to 12 weeks will be assessed using high-sensitivity C-reactive protein (hs-CRP) assay. Blood samples will be collected before dialysis sessions at baseline and after 12 weeks of treatment. The difference in CRP levels between the sertraline and placebo groups will be analyzed to determine the anti-inflammatory effect of sertraline in hemodialysis patients with depression.

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HAM-D) Score from Baseline to 12 Weeks | Baseline, Week 4, Week 8, and Week 12
  Depression severity will be measured using the Hamilton Depression Rating Scale (HAM-D), a validated tool for assessing depressive symptoms. HAM-D scores will be recorded at baseline, weeks 4, 8, and 12. The difference in scores between the sertraline and placebo groups will be evaluated to determine the antidepressant efficacy of sertraline.
Proportion of Patients Achieving a ≥50% Reduction in HAM-D Score | At Week 12
  The percentage of participants achieving a ≥50% reduction in HAM-D score from baseline to week 12 will be calculated. A higher proportion in the sertraline group compared to the placebo group will indicate better treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Irfan Jamil, Principal Investigator — Lahore General Hospital, Lahore
Locations (1):
- Nishtar Hospital, Multan, Multan, Punjab Province, Pakistan